CLINICAL TRIAL: NCT03535415
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone in Short Stature Children Due to Chronic Kidney Disease Before Transplantation
Brief Title: A Study to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone in Short Stature Children Due to Chronic Kidney Disease Before Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other); Beijing Children's Hospital (Other); Shanghai Children's Hospital (Other); Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Unknown); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Peking University First Hospital (Other); Fuzhou General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shengjing Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Tongji medical college huazhong university of science & technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci GH AQ CT-CKD
Record Dates: First submitted 2018-04-28; First posted 2018-05-24 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Dwarfism
MeSH Terms: conditions — Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhGH Injection (Experimental): rhGH 0.05mg/kg/d by subcutaneous injection
  Interventions: Drug: Recombinant Human Growth Hormone Injection (rhGH)
- Non-treatment control group (No Intervention): Only follow-up without treatment

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone Injection (rhGH) — rhGH 0.05mg/kg/d by subcutaneous injection
  Arms: rhGH Injection

SUMMARY:
This study aims to evaluate the efficacy and safety of recombinant human growth hormone injection in short stature children due to chronic kidney disease before transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent of the subjects or the legal guardian.
* Subjects and guardian are willing and able to cooperate to complete scheduled visits,treatment plans and laboratory tests and other procedures.
* Diagnosed as chronic kidney disease.
* Glomerular filtration rate (GFR) <75ml/per min/1.73m2.
* After the treatment and adjustment of hypertension, anemia, metabolic acidosis, malnutrition, renal osteopathy, hypothyroidism, etc..
* Chronological age: ≥2years and ≤14years.
* Height Standard Deviation Score(HtSDS) ≤-2SD for chronological age.
* Bone age: girls≤10 years; boys≤11years.
* Pre-pubertal (Tanner Stage I ) patients.
* No history of growth hormone treatment.

Exclusion Criteria:

* Subjects with abnormal liver functions.
* Subjects positive for anti-HBc, HbsAg or HbeAg in Hepatitis B virus tests.
* After adjustment heart function,Cardiac ejection fraction(EF) <50%.
* Subjects with highly allergic constitution or allergy to proteins or investigational product or its excipient.
* Subjects with systemic chronic disease or general infection or mental disease.
* Subjects with diabetes or impaired fasting glucose.
* Subjects with tumor or potential tumor.
* Subjects who are using glucocorticoid or immunosuppressant.
* Other causes for growth retardation.
* Inability to obtain accurate height measurements.
* Subjects who took part in other clinical trials within 3 months.
* Concomitant administration of other treatment that may have an effect on growth within 3 months.
* Other conditions which are unsuitable for this study in the opinion of the investigator.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The change of height standard deviation score of chronological age before and after treatment (ΔHT SDS) | 52 weeks，104 weeks

SECONDARY OUTCOMES:
Growth velocity | 12 months, 24 months
  365.25*（height at the time of assessment -height at baseline）/duration of treatment(days)
Bone maturation ( bone age/ chronological age: BA/CA) | 12 months, 24 months
IGF-1 (Insulin-like growth factor 1) SDS | 12 months, 24 months
IGF-1/IGFBP-3 molar ratio | 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (12):
- China (12):
  - Fuzhou general hospital of Nanjing military command, Fuzhou, Fujian
  - The first affiliated hospital of zhengzhou university, Zhengzhou, Henan
  - Tongji medical college huazhong university of science & technology, Wuhan, Hubei
  - Shengjing hospital of chian medical university, Shenyang, Liaoning
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Children's Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Children's hospital capital institute of pediatrics, Beijing
  - Peking university first hospital, Beijing
  - Children's hospital of Chongqing medical university, Chongqing
  - Children's Hospital of Fudan University, Shanghai
  - Children's Hospital of Shanghai, Shanghai